CLINICAL TRIAL: NCT00984048
Title: Prospective Study to Identify Molecular Mechanisms of Clinical Resistance to Standard First-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Study to Identify Mechanisms of Resistance to Standard Therapy in Patients With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Collaborators: Exactis Innovation (Other); Terry Fox Research Institute (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Gerald Batist, Principal Investigator, Jewish General Hospital
Other Study IDs: Q-CROC-01
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; FOLFOX; FOLFIRI; Avastin; Metastases; Liver; Colon cancer; Biomarkers; Resistance; Biobanking; Colorectal cancer with unresectable metastases to the liver
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue from a hepatic metastasis will be removed by needle core biopsy (NCB) obtained under radiologic guidance and will be flash-frozen. To obtain sufficient material for tissue banking, three needle core biopsies (NCB) will be removed from the same metastasis. Additionally, monthly whole blood samples will be collected, as well as plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FOLFOX, XELOX or FOLFIRI +/- bevacizumab: Patients are scheduled to receive first-line treatment for metastatic disease. They should be receiving at least one component of either FOLFOX, XELOX or FOLFIRI regimen with or without bevacizumab.
  Interventions: Other: Needle core biopsies of liver metastasis

INTERVENTIONS:
Other: Needle core biopsies of liver metastasis — No investigational products will be administered to subjects as part of this translational research study. A first-line chemotherapy regimen consisting of FOLFOX, XELOX or FOLFIRI +/- bevacizumab will be administered as per the standard of care at each treating institution. Needle core biopsies of liver metastasis will be collected and banked before the start of chemotherapy and at the time of progression. Additionally, blood samples will be drawn monthly and stored in the tissue biobank.

SUMMARY:
This is a multicenter translational study to understand therapeutic resistance in patients undergoing first-line chemotherapy (FOLFOX/Avastin, or FOLFIRI/Avastin) for metastatic colorectal cancer. Tissue samples from liver metastasis will be collected and banked before the start of chemotherapy and at the time of progression. Additionally, blood samples will be drawn monthly and stored in the tissue biobank.

DETAILED DESCRIPTION:
The major obstacle to the cure of cancer by pharmacological agents is resistance to these agents. Clinical responses of metastatic cancers to the most advanced chemotherapeutic agents usually range from 15 to 40%, indicating that intrinsic resistance, and acquired resistance occurs almost inevitably in those tumors that do respond. In patients with metastatic colorectal cancer, clinical resistance to a particular treatment is a clear endpoint (tumor growth), and is usually observed within 6-12 months of any given therapy. Thus, drug resistance and selecting appropriate therapeutic alternatives for drug-resistant cancer remain major dilemmas for oncologists.

The current first-line treatment for metastatic colorectal cancer in Quebec and much of North America is a combination called FOLFOX (the fluoro-pyrimidine 5-FU given as a 46-hour infusion, folinic acid and oxaliplatin) in combination with bevacizumab (Avastin®). An alternative regimen of cytotoxic drugs, also used with Avastin®, is FOLFIRI, which simply replaces oxaliplatin with the topoisomerase inhibitor irinotecan. In the metastatic setting, studies have not demonstrated significant differences between the two regimens, such that decision-making lacks definitive tools.

The objective of this study is to identify, in clinical samples, the molecular signature of clinically resistant colorectal cancer (CRC) patients for the most current and commonly used therapeutic agents. The goals of this study are two-fold. First, to build a biobank of blood and tissue specimens, prior to starting chemotherapy and at a determined time-point (progression of disease), from patients undergoing the same standard and well established first-line treatments (FOLFOX/bevacizumab or FOLFIRI/bevacizumab) for metastatic colorectal cancer. Second, to use state-of-the-art approaches by various collaborating laboratories to correlate clinical outcomes with molecular events that can be used to predict and circumscribe chemoresistance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically confirmed diagnosis of colorectal cancer, with at least one liver metastasis site available for biopsy.
2. For patients with liver only disease, patients deemed not to be initially resectable
3. Scheduled to receive first-line chemotherapy (FOLFOX/bevacizumab or FOLFIRI/bevacizumab) for metastatic disease.
4. Measurable metastatic disease (at least one unidimensionally measurable lesion) present after planned biopsy of metastatic site(s).
5. ECOG 0, 1 or 2.
6. Life expectancy of 12 or more weeks.
7. Age > 18 years.
8. Able to adhere to the study visit schedule and other protocol requirements.
9. Normal coagulation profile (PT, PTT, INR).

Exclusion Criteria:

1. Patients with initially resectable liver only metastases
2. Have received prior therapy for metastatic cancer. Prior adjuvant therapy is allowed.
3. Inadequate or unusable tissue as the only tissue available for biopsy.
4. Contraindication to any of the components of the the first-line chemotherapy regimen.
5. Known brain metastases or meningeal disease.
6. Female patients who are pregnant or breastfeeding.
7. Concurrent treatment with other anti-cancer therapy (palliative radiation is allowed but patients must have a metastatic site available for re-biopsy that has not been irradiated).
8. Abnormal coagulation profile, any anti-coagulant therapy.
9. Known infection with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients with a confirmed diagnosis of colorectal cancer with the presence of liver metastasis, who will be receiving first-line treatment (FOLFOX/bevacizumab or FOLFIRI/bevacizumab) for metastatic disease.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2009-08; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Changes in biomarkers in patients that have acquired clinical resistance. | 4 years
  Liver needle core biopsies are obtained pre-treatment and at progression of disease from all patients. These are used to discover exploratory biomarkers of resistance to FOLFOX/bevacizumab and FOLFIRI/bevacizumab

SECONDARY OUTCOMES:
Number of participants with adverse events relating to the liver biopsy procedure | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, MD, Study Director — Jewish General Hospital, Segal Cancer Center
Locations (15):
- University Hospital Leuven, Leuven, Belgium
- Canada (14):
  - The Moncton Hospital, Moncton, New Brunswick
  - Dr. Georges L. Dumont University Hospital, Moncton, New Brunswick
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital Notre-Dame, Montreal, Quebec
  - Hôpital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St-Mary's Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital Sacré-Coeur, Montreal, Quebec
  - Hôtel-Dieu du Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided